CLINICAL TRIAL: NCT06221995
Title: Energy Requirements in Patients With Ulcerative Colitis Undergoing Total Rectocolectomy and Ileoanal Anastomosis J-pouch
Brief Title: Energy Expenditure in Patients With Ulcerative Colitis Undergoing Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Evangelismos Hospital (Other)
Responsible Party: Principal Investigator, Dimitrios Karayiannis, Director, Department of Clinical Nutrition, Evaggelismos General Hospital, Athens, Evangelismos Hospital
Other Study IDs: PouchEH
Record Dates: First submitted 2024-01-02; First posted 2024-01-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis; Surgery
Keywords: Ulcerative Colitis; energy requirements; ileoanal anastomosis; j-pouch
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ulcerative Colitis patients undergoing proctocolectomy: Measurement of resting energy expenditure among patients with Ulcerative Colitis about to undergo proctocolectomy with ileoanal j-pouch anastomosis
  Interventions: Diagnostic Test: Indirect Calorimetry

INTERVENTIONS:
Diagnostic Test: Indirect Calorimetry — Resting energy expenditure measurement
  Other Names: Resting energy expenditure measurement

SUMMARY:
A prospective observational study to assess the energy needs of Ulcerative Colitis patients undergoing total proctocolectomy with ileoanal j-pouch anastomosis.

DETAILED DESCRIPTION:
Total proctocolectomy with creation of ileoanal j-pouch anastomosis is the gold-standard surgical procedure for familial polyposis, for ulcerative colitis unresponsive to medication and for colitis associated with dysplasia requiring total colectomy.

Patients postoperatively face difficulties in maintaining their physical condition and quality of life due to potential complications such as surgical, mechanical, inflammatory and functional disorders increasing the rates of malnutrition. Postoperative changes as regards anthropometric characteristics and nutritional status have not been fully elucidated.

Therefore, the need arises to calculate the energy needs of patients with ileoanal j-pouch anastomosis, given the lack of corresponding data and the possible differentiation of energy needs from a similar group of patients undergoing colorectal surgery.

Of particular interest is the body composition of ileoanal anastomosis patients, which has been studied very little ), and the extent to which their energy needs are met, given dietary restrictions both preoperatively and postoperatively.

It is therefore necessary to determine the energy needs, as well as the degree of their coverage by the diet, of UC patients undergoing proctocolectomy with creation of ileoanal j-pouch anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ulcerative colitis and planned proctocolectomy with ileoanal j-pouch anastomosis surgery or patients who are to undergo subtotal colectomy.
* Age over 18 years.
* Written informed consent to take part in the study.
* Speaking ability in Greek or English.
* Able to get tested fasted;

Exclusion Criteria:

* Age under 18 years.
* Existence of pregnancy.
* Inability to breathe inside the indirect calorimetry mask for the time required for the measurement.
* Use of medications that may affect body metabolism will be evaluated individually (e.g. cortico-steroids etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Ulcerative Colitis about to undergo proctocolectomy with ileoanal j-pouch anastomosis. As control group, it is planned to enroll patients about to undergo subtotal colectomy, matched with the patient group in terms of gender, age and body mass index.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Amount of resting energy expenditure (kcal/day) | Before surgery, 1 week postoperatively, 3 months postoperatively
  To evaluate total energy needs of patients who undergo proctocolectomy with ileoanal j-pouch

SECONDARY OUTCOMES:
IBDQ | Before surgery and 1 week after Surgery
  Inflammatory Bowel Disease Questionnaires (IBDQ), a widely used questionnaire for HRQoL assessment in patients with inflammatory bowel diseases (IBDs)
Resting energy expenditure change (kcal/day) | 1 week postoperatively and 3 months postoperatively
  Changes in daily energy expenditure after surgery compared to pre surgery assesment.
Bristol stool form scale, min: type 1 (hard solid stools, better outcome) - max: type 7 (liquid stools, worst outcome) | Before surgery, 1 week postoperatively, 6 months after surgery
  Longitudinal changes in Bristol stool form scale score before and after surgery.
Post operative weight loss | 1 week postoperatively, 3 months postoperatively
  Post operative weight loss will be assessed by measuring the post weight on the date of surgery and adjusting for the baseline weight in kg.
Post operative Energy intake. | 1 week postoperatively, 3 months postoperatively
  Total energy intake measured in calories after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Karagiannis, Dr, Study Director — Evangelismos General Hospital of Athens
Locations (1):
- Evangelismos General Hospital of Athens, Athens, Attica, Greece